CLINICAL TRIAL: NCT02911909
Title: Moderated Blood Flow Restriction After Anterior Cruciate Ligament
Brief Title: Moderated Blood Flow Restriction After Anterior Cruciate Ligament Reconstruction
Acronym: Delfi
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment was unsuccessful
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, James Cook, William & Kathryn Allen Distinguished Professor in Orthopaedic Surgery, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2004255
Record Dates: First submitted 2016-08-05; First posted 2016-09-22 (Estimated); Results first posted 2020-03-11 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Anterior Cruciate Ligament Tear
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Standard rehabilitation (Active Comparator): Patients will receive standard post-operative ACL rehabilitation
  Interventions: Other: Standard rehabilitation
- Delfi moderated blood flow restriction (Experimental): Patients will receive Delfi moderated blood flow post-operative ACL rehabilitation
  Interventions: Device: Delfi

INTERVENTIONS:
Device: Delfi — Patients will receive standard of care post-operative ACL reconstruction rehabilitation plus the Delfi moderated blood flow restriction therapy.
  Other Names: moderated blood flow restriction device
  Arms: Delfi moderated blood flow restriction
Other: Standard rehabilitation — Patients will receive standard of care post-operative ACL reconstruction rehabilitation
  Arms: Standard rehabilitation

SUMMARY:
The aim of this study is to determine if there is a difference in post operative rehabilitation after anterior cruciate ligament (ACL) reconstruction surgery while using moderated blood flow therapy vs. standard physical therapy. All patients undergoing ACL reconstruction, between the ages of 18-30, that consent to taking part in the study, and meet eligibility criteria, will be included in the study. Patients will be followed for two years to determine any differences in muscle strength, thigh circumference, knee range of motion, pain, functional and activity levels, patient satisfaction, levels of Human growth hormone HGH), Insulin-like Growth Factor (IGF), and Creatine Kinase (CK), KT2000, and Lachman physical examination.

DETAILED DESCRIPTION:
The study will be a prospective, randomized, controlled trial between two treatment cohorts. A total of 50 patients will be enrolled in the study. Informed consent will be obtained in clinic prior to any surgical intervention, per the IRB protocol. Enrollees will receive a copy of the consent and HIPAA form. All patients that meet inclusion criteria who consent to participate in the study will then be randomly assigned to either the control group or moderated blood flow therapy group. Randomization will occur by autogenerated permutated 1:1 block randomization using electronic assignment from the orthopaedic research team prior to initiation of post-operative therapy. The control group will undergo standard of care, post-operative ACL reconstruction rehabilitation. The treatment group will also receive standard ACL rehabilitation combined with Delfi moderated blood flow restriction therapy. Patients will follow up at standard of care clinic visits and participate in the same standard of care physical therapy protocol for ACL reconstruction. Baseline measurements of thigh circumference, knee ROM, KT 2000, Lachman exam, and labs for HGH, IGF, and CK will be obtained preoperatively. Patients will also complete preoperative IKDC, Tegner, PROMIS, and VAS pain surveys. Measurements of thigh circumference and knee range of motion will occur at 2 week intervals post operatively. Strength testing will start at 6 weeks post-operatively. These measurements will occur during standard therapy sessions. KT 2000 and Lachman exam will be performed at 4, 6, 8, and 12 months post operatively. A standard functional return to sport evaluation will be performed at the 4, 6, 8, and 12 month postoperative visits. Labs for HGH, IGF, and CK will be drawn at 2, 6, 12, and 24 weeks. VAS pain scores will be recorded before and after each therapy session. The PROMIS, IKDC, and Tegner surveys will be given at 4, 6, 8, 12 month intervals. The study will conclude at 12 month follow up. All post-operative visits will be standard of care. No additional clinic visits will be required for this study. Background patient information will be collected including age, sex, BMI, and co-morbidities.

The control group will be necessary to provide a baseline measure on which moderated blood flow therapy will be compared.

Blinding of the subject will not be possible as the patient will be able to recognize if they have or have not had the moderated blood flow (Delfi) device applied during therapy and application of a sham-device is not practical or considered standard of care. Evaluators performing measurements will be blinded to the patient's treatment group during assessment of muscle strength, thigh circumference, knee range of motion, Lachman exam, and KT2000. Surgeons will also be blinded to the respective treatment groups. All other outcome measures are objective and quantitative.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18-30 years of age.
* Diagnosis of isolated anterior cruciate ligament (ACL) tear and pending ACL reconstruction.

Exclusion Criteria:

* age <18 years old or >30 years old
* Multi-ligament knee injury
* Revision ACL reconstruction
* History or peripheral vascular disease
* History of deep vein thrombosis or pulmonary embolism
* Any contraindication to moderated blood flow restriction therapy
* Inability to comply with post-operative ACL reconstruction rehabilitation
* If meniscal repair or a cartilage procedure is performed at the time of surgery that would preclude the patient from being able to follow the standard post-operative ACL rehabilitation.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-10-21 (Actual); Study Completion 2019-10-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Cook, Principal Investigator — University of MO-Columbia
Locations (1):
- Missouri Orthopaedic Institute, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Rehabilitation | Delfi Moderated Blood Flow Restriction
Started | 4 | 3
Completed | 2 | 0 (No Data was obtained in the study group.)
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Population: of the 3 patients in the delfi group, 1 did not undergo surgery after consent. For the other 2, our Physical Therapy department was unable to perform the required preoperative evaluation. No data was obtained in the Delfi Group
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Rehabilitation | Delfi Moderated Blood Flow Restriction | Total
Number analyzed (Participants) | 2 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.5 (1.5) |  | 29.5 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  | 1
  Male | 1 |  | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 2 |  | 2
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Muscle Strength
Description: Compare mean peak muscle strength at 60 degrees of knee flexion (during extension) of the involved leg between the blood restriction and the control groups
Time Frame: 12 months
Population: No Subjects in the Deflfi group completed the muscle strength evaluation at 12 months
Measure: Mean (Standard Deviation); unit: FT-LBS
Arm/Group | Standard Rehabilitation | Delfi Moderated Blood Flow Restriction
Number analyzed (Participants) | 2 | 0
FT-LBS | 95.5 (60.7) |

2. Secondary Outcome: Range of Motion
Description: Compare the total Range of motion of the involved leg at 12 months between the Delfi and the control group
Time Frame: 12 months
Population: No patient in the Delfi group complete the 12 months evaluation / No data obtained in the Delfi group
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Standard Rehabilitation | Delfi Moderated Blood Flow Restriction
Number analyzed (Participants) | 2 | 0
Degrees | 135 (5) |

3. Secondary Outcome: Tegner Activity Survey Score
Description: Compare the Tegner Activity Survey score mean between the Delfi and the control group.
  Tegner activity level scale is a scale that aims to provide a standardized method of grading work and sporting activities. Tegner activity level scale is a graduated list of activities of daily living, recreation, and competitive sports. The patient is asked to select the level of participation that best describes their current level of activity and that before injury. The score varies from 0-10. A score of 0 represents sick leave or disability pension because of knee problems, whereas a score of 10 corresponds to participation in national and international elite competitive sports >6 score can only be achieved if the person participates in recreational or competitive sport.
Time Frame: 12 months
Population: No patient in the Delfi group complete the 12 months evaluation / No data obtained in the Delfi group
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Rehabilitation | Delfi Moderated Blood Flow Restriction
Number analyzed (Participants) | 2 | 0
score on a scale | 1 (1) |

4. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) Survey Score.
Description: Compare the mean Patient-Reported Outcomes Measurement Information System Global Physical health row score (PROMIS) between the Delfi and the control group.
  PROMIS® (Patient-Reported Outcomes Measurement Information System) is a set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children. It can be used with the general population and with individuals living with chronic conditions. The Score is represented in a 0 to 100 scale. Zero is the worst possible outcome and 100 is teh best possible outcome
Time Frame: 12 months
Population: No patient in the Delfi group complete the 12 months evaluation / No data obtained in the Delfi group
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Rehabilitation | Delfi Moderated Blood Flow Restriction
Number analyzed (Participants) | 2 | 0
score on a scale | 11.5 (1.5) |

5. Secondary Outcome: International Knee Documentation Committee (IKDC) Survey Score
Description: Compare the mean International Knee Documentation Committee (IKDC) survey score between the delfi and the control group The IKDC Questionnaire is a subjective scale that provides patients with an overall function score. The questionnaire looks at 3 categories: symptoms, sports activity, and knee function. The symptoms subscale helps to evaluate things such as pain, stiffness, swelling and giving-way of the knee. Meanwhile, the sports activity subscale focuses on functions like going up and down the stairs, rising from a chair, squatting and jumping. The knee function subscale asks patients one simple question: how is their knee at present versus how was their knee prior to injury?
  Scores are obtained by summing the individual items, then transforming the crude total to a scaled number that ranges from 0 to 100. This final number is interpreted as a measure of function with higher scores representing higher levels of function.
Time Frame: 12 months
Population: No patient in the Delfi group complete the 12 months evaluation / No data obtained in the Delfi group
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Rehabilitation | Delfi Moderated Blood Flow Restriction
Number analyzed (Participants) | 2 | 0
score on a scale | 72.415 (27.585) |

6. Secondary Outcome: Visual Analog Scale (VAS)
Description: Compare the mean VAS scores (0 no pain - 10 worse pain ever) between the Delfi and the control group
Time Frame: 12 months
Population: No patient in the Delfi group complete the 12 months evaluation / No data obtained in the Delfi group
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Rehabilitation | Delfi Moderated Blood Flow Restriction
Number analyzed (Participants) | 2 | 0
score on a scale | 1.5 (1.5) |

7. Secondary Outcome: Tight Circumference
Description: Compare tight circumference of the involved leg between Delfi and the control group
Time Frame: 12 months
Population: No patient in the Delfi group complete the 12 months evaluation / No data obtained in the Delfi group
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Standard Rehabilitation | Delfi Moderated Blood Flow Restriction
Number analyzed (Participants) | 2 | 0
cm | 49.375 (0.625) |

8. Secondary Outcome: KT-2000 Anterior Tibial Translation
Description: Compare the mean anterior translation of the tibia between delfi and control groups anterior translation was measured using a KT-2000 device
Time Frame: 12 months
Population: No patient in the Delfi group complete the 12 months evaluation / No data obtained in the Delfi group
Measure: Mean (Standard Deviation); unit: milimiters
Arm/Group | Standard Rehabilitation | Delfi Moderated Blood Flow Restriction
Number analyzed (Participants) | 2 | 0
milimiters | 9 (1) |

9. Secondary Outcome: CK Level
Description: Compare CK levels at 12 months between delfi and control group
Time Frame: 12 months
Population: Samples were not processed due to study termination
Arm/Group | Standard Rehabilitation | Delfi Moderated Blood Flow Restriction
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: HGH Level
Description: Compare mean HGH blood levels between the delfi and the control group
Time Frame: 12 months
Population: Samples were not processed due to study termination
Arm/Group | Standard Rehabilitation | Delfi Moderated Blood Flow Restriction
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: IGF Level
Description: Compare the mean IGF blood values between delfi and control group
Time Frame: 12 months
Population: samples were not processed due to study termination
Arm/Group | Standard Rehabilitation | Delfi Moderated Blood Flow Restriction
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: Adverse events: 0
Arm/Group | Standard Rehabilitation | Delfi Moderated Blood Flow Restriction
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/0
Other Adverse Events (participants affected / at risk) | 0/2 | 0/0

LIMITATIONS AND CAVEATS:
Finding patients that meet all the inclusion criteria was cumbersome. Some patients after enrollment had intra-operative findings that would later make them not eligible to keep participating in the study (required procedures beyond ACL recon)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-14): https://cdn.clinicaltrials.gov/large-docs/09/NCT02911909/Prot_SAP_000.pdf